CLINICAL TRIAL: NCT01097057
Title: Mobilization of Autologous Peripheral Blood Stem Cells (PBSC) in CD20+ Lymphoma Patients Using RICE, G-CSF (Granulocyte-Colony Stimulating Factor), and Plerixafor
Brief Title: Rituximab, Combination Chemotherapy, Filgrastim (G-CSF), and Plerixafor in Treating Patients With Non-Hodgkin Lymphoma Undergoing Mobilization of Autologous Peripheral Blood Stem Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leona Holmberg, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2310.00; NCI-2009-01562 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2310.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Carboplatin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Ifosfamide; Leukapheresis; plerixafor; ferric pyrophosphate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (rituximab, etoposide, carboplatin, ifosfamide) (Experimental): Patients receive rituximab IV on day 1, etoposide IV on days 2-4, carboplatin IV on day 3, and ifosfamide IV on day 3 over 24 hours. Patients also receive G-CSF SC once daily beginning on day 6 and continuing until apheresis is completed and plerixafor SC once daily for up to 4 days beginning 24 hours after recovery from nadir and continuing until apheresis is completed. Patients may undergo up to 4 apheresis procedures until the optimal number of CD34+ cells are collected.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Biological: Filgrastim; Drug: Ifosfamide; Procedure: Leukapheresis; Drug: Plerixafor; Biological: Rituximab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Procedure: Leukapheresis — Given through catheter
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Drug: Plerixafor — Given SC
  Other Names: AMD 3100; JM-3100; Mozobil; SDZ SID 791
Biological: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar BI 695500; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; RTXM83

SUMMARY:
This phase II trial is studying how well giving rituximab; ifosfamide, carboplatin, and etoposide (ICE) combination chemotherapy; and filgrastim (G-CSF) together with plerixafor works in treating patients with non-Hodgkin lymphoma undergoing mobilization of autologous peripheral blood stem cells. Giving chemotherapy (ICE) with monoclonal antibodies, such as rituximab, stops the growth of cancer cells by stopping them from dividing or by killing them and helps get better autologous stem cell product. Giving colony-stimulating factors, such as G-CSF, and plerixafor helps stem cells move from the patient's bone marrow to the blood so they can be collected and stored for future autologous transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the efficacy of combining RICE (rituximab-ifosfamide-carboplatin-etoposide regimen [R-ICE regimen]), G-CSF, and plerixafor to collect autologous peripheral blood stem cell (PBSC) for non-Hodgkin's lymphoma (NHL) patients by: the number of days of apheresis required to reach >= 5 x 10^6 cluster of differentiation (CD)34 cells/kg and by the total number of CD34 cells/kg collected in a maximum of 4 days if >= 5 x 10^6 CD34 cells/kg is not obtained.

OUTLINE:

Patients receive rituximab intravenously (IV) on day 1, etoposide IV on days 2-4, carboplatin IV on day 3, and ifosfamide IV on day 3 over 24 hours. Patients also receive filgrastim subcutaneously (SC) once daily beginning on day 6 and continuing until apheresis is completed and plerixafor SC once daily for up to 4 days beginning 24 hours after recovery from nadir and continuing until apheresis is completed. Patients may undergo up to 4 apheresis procedures until the optimal number of CD34+ cells are collected.

After completion of study treatment, patients are followed up at 30 days and then periodically for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD20+ non-Hodgkin's lymphoma
* Left ventricular ejection fraction at rest >= 50% demonstrated by multi gated acquisition scan (MUGA) or echocardiogram
* Bilirubin =< 2.0 mg/dL (except for isolated hyperbilirubinemia attributed to Gilbert syndrome)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 times the upper limit of normal
* Creatinine clearance (calculated creatinine clearance is permitted) > 50 mL/min
* Signed informed consent
* Planned autologous transplant within 3 months after collection of peripheral blood stem cells (PBSCs)

Exclusion Criteria:

* Karnofsky performance score < 70%
* Uncontrolled bacterial, viral, or fungal infection (currently taking medication and with progression or no clinical improvement)
* Prior other malignancies except resected basal cell carcinoma or treated cervical carcinoma or breast cancer in situ; cancer treated with curative intent > 5 years previously will be allowed
* Pregnant or breastfeeding
* Fertile men or women unwilling to use contraceptive techniques from the time of chemo-mobilization
* Prior autologous or allogeneic hematopoietic stem cell transplant (HSCT)
* Human immunodeficiency virus (HIV) positive
* Plan to be treated on another investigational therapy within 4 weeks of enrolling on this study
* Hepatitis B carriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11-09 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2017-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Rituximab, Etoposide, Carboplatin, Ifosfamide)
Started | 20
Completed | 17
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Rituximab, Etoposide, Carboplatin, Ifosfamide)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: Years] | 66 [42 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients to Mobilize ≥5 x 10^6 CD34 Cells/kg Autologous PBSC (Efficacy)
Description: Number of patients who achieved ≥5 x 10^6 CD34 cells/kg autologous PBSC collection by apheresis.
Time Frame: One Month
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab, Etoposide, Carboplatin, Ifosfamide)
Number analyzed (Participants) | 17
Participants | 17

2. Primary Outcome: Number of Patients Who Achieved ≥5 x 10^6 CD34 Cells/kg in ≤4 Apheresis Days
Description: Number of patients to collect at least 5 x 10^6 CD34 cells/kg in under 4 apheresis procedures.
Time Frame: Up to Four Apheresis Days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab, Etoposide, Carboplatin, Ifosfamide)
Number analyzed (Participants) | 17
Participants | 17

3. Primary Outcome: Number of Participants Requiring One or Two Apheresis Collection Days to Reach ≥5 x 10^6 CD34 Cells/kg
Description: Number of participants requiring one or two apheresis collection days to reach collection goal.
Time Frame: Up to Four Apheresis Days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab, Etoposide, Carboplatin, Ifosfamide)
Number analyzed (Participants) | 17
Participants
  One apheresis collection day | 15
  Two apheresis collection days | 2
  Three apheresis collection days | 0
  Four apheresis collection days | 0

4. Primary Outcome: Total Number of Participants Who Did Not Collect ≥5 x 10^6 CD34 Cells/kg in a Maximum of Four Apheresis Days
Description: Number of participants who did not collect ≥5 x 10^6 CD34 cells/kg in up to four apheresis days
Time Frame: Up to Four Apheresis Days
Population: Note: No patients were in this category.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab, Etoposide, Carboplatin, Ifosfamide)
Number analyzed (Participants) | 17
Participants | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Rituximab, Etoposide, Carboplatin, Ifosfamide)
All-Cause Mortality (participants affected / at risk) | 5/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Rituximab, Etoposide, Carboplatin, Ifosfamide) (N=20)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 — No treatment related deaths
Atrial Fibrillation (Cardiac disorders) | 1 — No treatment related deaths
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Rituximab, Etoposide, Carboplatin, Ifosfamide) (N=20)
DVT (Vascular disorders) | 1 — Non-hematological toxicity. Grading of toxicity according NCI-CTCAE version 3. Asymptomatic line-associated DVT requiring therapeutic anticoagulant.
Cellulitis (Infections and infestations) | 1 — Non-hematological toxicity. Grading of toxicity according NCI-CTCAE version 3. Cellulitis at Hickman site
Hyperglycemia (Metabolism and nutrition disorders) | 2 — Non-hematological toxicity. Grading of toxicity according NCI-CTCAE version 3. One patient had both hyperglycemia and cellulitis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No